CLINICAL TRIAL: NCT02234804
Title: The Does Optical Coherence Tomography Optimize Revascularization (DOCTOR) Recross Study
Acronym: DOCTOR Recross
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Abbott Medical Devices (Industry); Medtronic (Industry)
Responsible Party: Principal Investigator, Niels Ramsing Holm, MD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-111-13
Record Dates: First submitted 2014-06-05; First posted 2014-09-09 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Disease
Keywords: Coronary angiography (CAG); Percutaneous coronary intervention (PCI); OCT; Stent
MeSH Terms: conditions — Coronary Disease | interventions — Stents; Cerebral Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Medtronic Resolute Integrity stent (Experimental): Comparing Medtronic Resolute Integrity and Xience Prime for stent strut apposition in the SB ostium
  Interventions: Procedure: Angiography; Procedure: OCT
- OCT (Experimental): OCT to guide wire recrossing and reduce stent strut malapposition after kissing balloon dilatation.
  Interventions: Device: Xience Prime Stent; Device: Medtronic Resolute Integrity stent
- Angiography (Active Comparator): Angiography to guide wire recrossing and reduce stent strut malapposition after kissing balloon dilatation.
  Interventions: Device: Xience Prime Stent; Device: Medtronic Resolute Integrity stent
- Xience Prime stent (Active Comparator): Comparing Medtronic Resolute Integrity and Xience Prime for stent strut apposition in the SB ostium
  Interventions: Procedure: Angiography; Procedure: OCT

INTERVENTIONS:
Device: Xience Prime Stent
  Other Names: Stent
  Arms: Angiography; OCT
Device: Medtronic Resolute Integrity stent
  Other Names: Stent
  Arms: Angiography; OCT
Procedure: Angiography
  Other Names: CAG
  Arms: Medtronic Resolute Integrity stent; Xience Prime stent
Procedure: OCT
  Arms: Medtronic Resolute Integrity stent; Xience Prime stent

SUMMARY:
Prospective, controlled, double randomized, non-blinded, multicenter, investigator initiated, academic superiority trial comparing optical coherence tomography (OCT) guided vs. angiography guided wire recrossing in jailed side branches (SB) (1. randomization 1:1)(superiority) and comparing Medtronic Resolute Integrity and Xience Prime for stent strut apposition in the SB ostium (2. randomization 1:1) (superiority). Acute primary endpoint and 30 days clinical follow-up.

Hypothesis: OCT guided wire recrossing in bifurcation stenting results in less malapposed struts in the segment facing the SB ostium.

Secondary hypothesis: Treatment by Medtronic Resolute Integrity stent results in less malapposed struts at the bifurcation segment compared to treatment by the Abbott Xience Prime stent.

DETAILED DESCRIPTION:
Purpose:

To assess the ability of OCT to guide wire recrossing and reduce stent strut malapposition after kissing balloon dilatation.

To compare stent strut apposition after treatment by two different stent designs using both guiding strategies of wire recrossing.

ELIGIBILITY:
Inclusion Criteria:

* Stable or unstable angina pectoris or silent angina pectoris.
* De novo coronary bifurcation lesions at "LAD/diagonal", "Cx/obtuse marginal", "right coronary artery (RCA)- posterior descending artery (PDA)/posterolateral branch" or "left main (LM)/Cx/LAD".
* All Medina classes except Medina 0.0.1.
* Diameter of side branch ≥2.5 mm.
* Diameter stenosis >50% by operator's visual assessment
* Signed informed consent

Exclusion Criteria:

* ST-elevation infarction within 48 hours.
* Side branch lesion length >5 mm.
* Expected survival < 1 year
* Severe heart failure (NYHA≥III)
* S-creatinine >120 µmol/l.
* Allergy to Contrast media, Aspirin, Clopidogrel, Ticagrelor, Ticlopidine, Everolimus or Zotarolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Cross sectional stent strut malapposition in the main vessel bifurcation segment facing the side-branch ostium compared for optical coherence tomography and angioguided recrossing strategy | Baseline

SECONDARY OUTCOMES:
Procedural: 1. Success in recrossing into designated strut hole when visible and indicated | Baseline
Procedural: 2. Procedure duration (sheath insertion to closure device excluding treatment of other vessels) | Baseline
Procedural: 3. Contrast use | Baseline
Procedural: 4. Fluoroscopy time | Baseline
Optical coherence tomography endpoints: 5. Malapposition in the main vessel segment limited by and facing the side-branch ostium compared for stent type (second randomization) | Baseline
Optical coherence tomography endpoints: Malapposition in the proximal and distal main vessel segments and in the quadrants opposite to the side branch origin for stent type and recross strategy | Baseline
Optical coherence tomography endpoints: Distance between malapposed strut and vessel wall in all segments for stent type and recross strategy | Baseline
Optical coherence tomography endpoints: Minimum expansion of the stents expressed as absolute area and percentage of the closest reference area, for stent type and recross strategy | Baseline
Optical coherence tomography endpoints: Ostial stent area stenosis by optical coherence tomography (side branch reference area by 3D QCA) | Baseline
Angiographic endpoints: Segmental assessment; Proximal edge, proximal main vessel, bifurcation segment, distal main vessel, distal edge, ostial 5 mm of side branch. Pre and post side branch intervention | Baseline
Ostial side branch area stenosis | Baseline
Ostial side branch acute gain after main vessel (MV) stenting | Baseline
Minimal luminal area of all segments | Baseline
Angiographic area stenosis of all other segments | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Niels R Holm, MD, Principal Investigator — Aarhus University Hospital Skejby
Locations (3):
- University Hospitals Leuven, Leuven, Belgium
- Aarhus University Hspital, Aarhus N, Denmark
- Royal Brompton Hospital, London, United Kingdom